CLINICAL TRIAL: NCT00563940
Title: Short-term Effects of Intravitreal Bevacizumab and Triamcinolone in Patients With Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: AUG 044/07; KEK E: 29-03-07
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; OCT

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
Diabetic macular edema is a common complication of ocular diabetes mellitus and can cause blindness. Hypoxygenation of the retina stimulates tissue mediators, especially different subtypes of vascular endothelial growth factor (VEGF). VEGF is responsible for proliferation, extension and increased permeability of the vessels. The aim of our study was to examine the short-term effect of intravitreal bevacizumab (Avastin® 1.25 mg in 0.05 ml) and triamcinolone on visual acuity and central retinal thickness in patients with clinically significant diabetic macular edema (CSME).

ELIGIBILITY:
Inclusion Criteria:

* clinical significant macular edema

Exclusion Criteria:

* retinal thickness < 250 µm

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical significant macular edema
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Central retinal thickness | 4, 8, 12, 24, 72, and 168 hours

SECONDARY OUTCOMES:
BCVA | 4, 8, 12, 24, 72, and 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ute Wolf-Schnurrbusch, MD, Principal Investigator — University of Bern; Sebastian Wolf, MD PhD, Study Director — University of Bern
Locations (1):
- Klinik und Poliklinik für Augenheilkunde, Bern, Switzerland